CLINICAL TRIAL: NCT04565444
Title: The Effects of Acute Nutritional Ketosis on Myofibrillar Protein Synthesis in Young Men
Brief Title: Ketones and Muscle Protein Synthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Tyler Churchward-Venne, Tyler A. Churchward-Venne, Ph.D., Assistant Professor, McGill University, McGill University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A11-M51-19A
Record Dates: First submitted 2020-09-17; First posted 2020-09-25 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Ketosis; Regulation of Muscle Protein Synthesis
Keywords: ketone; protein metabolism; muscle
MeSH Terms: conditions — Ketosis | interventions — Ketones; Proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ketone (Experimental): Ketone monoester supplement (R)-3-hydroxybutyl (R)-3-hydroxybutyrate based on participants' body weight (0.36g/kg body weight) and carbohydrate control.
  Interventions: Dietary Supplement: Ketone
- Ketone + Protein (Experimental): Ketone monoester supplement (R)-3-hydroxybutyl (R)-3-hydroxybutyrate based on participants' body weight (0.36g/kg body weight) and 10g of whey protein.
  Interventions: Dietary Supplement: Ketone + Protein
- Protein (Experimental): Carbohydrate control and 10g of whey protein.
  Interventions: Dietary Supplement: Protein

INTERVENTIONS:
Dietary Supplement: Ketone — * Ketone monoester supplement (R)-3-hydroxybutyl (R)-3-hydroxybutyrate based on participants' body weight (0.36g/kg body weight)
  * Isocaloric carbohydrate control: dextrose + vanilla flavouring
  Arms: Ketone
Dietary Supplement: Ketone + Protein — * Ketone monoester supplement (R)-3-hydroxybutyl (R)-3-hydroxybutyrate based on participants' body weight (0.36g/kg body weight)
  * 10g Whey Protein
  * L-[ring-2H5]-phenylalanine tracer (enriched to 4%)
  Arms: Ketone + Protein
Dietary Supplement: Protein — * Isocaloric carbohydrate control: dextrose + stevia
  * 10g Whey Protein
  * L-[ring-2H5]-phenylalanine tracer (enriched to 4%)
  Arms: Protein

SUMMARY:
Ketones are natural substances normally produced by the body during prolonged fasting and starvation, or in response to a "ketogenic" diet to be used as fuel by the brain and muscles. Ketones are therefore similar to dietary proteins, carbohydrates and fats since they represent a source of energy for the body. In addition to serving as a source of energy, ketones have also been shown to stimulate increased rates of muscle protein synthesis in humans.

The ingestion of dietary protein is well established to stimulate an increase in the rate of protein synthesis in skeletal muscle. The rate of muscle protein synthesis can be maximized following the intake of 20g of protein. As a result, smaller doses of protein (i.e. 10g) represent a sub-optimal dose of protein because there is still room for improvement concerning muscle protein synthesis.

Recently ketone-containing food products have become available that elevate ketone levels in the body without the need for ketogenic diets or prolonged fasting. Therefore, the purpose of this study is to measure skeletal muscle protein synthesis rates after ingesting the following:

1. Ketone monoester
2. Ketone monoester supplemented with sub-optimal dose of whey protein
3. Sub-optimal dose of whey protein

It is hypothesized that muscle protein synthesis rates will increase following the ingestion of a ketone-containing beverage. Further, muscle protein synthesis rates will be enhanced when the ketone-containing beverage and sub-optimal protein dose are taken together.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged between 18-35 years inclusive
* Healthy, moderately active
* BMI < 30 kg/m2 and > 18.5 kg/m2
* Having given informed consent

Exclusion Criteria:

* Presence of any identified metabolic or intestinal disorders
* Use of tobacco products
* Allergies to milk proteins (whey or casein)
* Lactose intolerance
* Phenylketonuria (PKU)
* A history of neuromuscular problems
* Previous participation in amino acid tracer studies
* Adherence to a strict vegetarian or vegan diet
* Current use of ketone supplements or adherence to a ketogenic diet
* Use of medications known to affect protein metabolism
* Diagnosis of Diabetes
* Engagement in sports or physical exercise 5 or more days per week

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
Fractional synthetic rate of muscle protein synthesis (myofibrillar) | 0-5 hours in the post-prandial period

SECONDARY OUTCOMES:
Fractional synthetic rate of muscle protein synthesis (myofibrillar) | 0-3 hours in the pre-prandial period; 0-2 hours, and 2-5 hours into the post-prandial period
Plasma enrichments (in moles percent excess) of L-[ring-2H5]-phenylalanine | 3 hours pre-prandial to 5 hours post-prandial
Plasma glucose concentration (mmol/L) | 3 hours pre-prandial to 5 hours post-prandial
Plasma insulin concentration (pmol/L) | 3 hours pre-prandial to 5 hours post-prandial
Plasma amino acid concentrations (mmol/L) | 3 hours pre-prandial to 5 hours post-prandial
Capillary blood Beta-OHB concentrations (mmol/L) | 0-5 hours in the post-prandial period
Signaling molecule phosphorylation status | 0, 2, and 5 hours into the post-prandial period
  The use of Western blots to measure the phosphorylation status of signaling molecules involved in protein synthesis ie. mTOR, p70S6k, 4E-BP1

CONTACTS AND LOCATIONS:
Overall Officials: Tyler A Churchward-Venne, Ph.D., Principal Investigator — McGill University
Locations (1):
- Exercise Metabolism and Nutrition Research Laboratory, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Hannaian SJ, Lov J, Hawley SE, Dargegen M, Malenda D, Gritsas A, Gouspillou G, Morais JA, Churchward-Venne TA. Acute ingestion of a ketone monoester, whey protein, or their co-ingestion in the overnight postabsorptive state elicit a similar stimulation of myofibrillar protein synthesis rates in young males: a double-blind randomized trial. Am J Clin Nutr. 2024 Mar;119(3):716-729. doi: 10.1016/j.ajcnut.2024.01.004. Epub 2024 Jan 11. PMID 38215886